CLINICAL TRIAL: NCT01924104
Title: Effects of Low Dose Aspirin and Low Molecular Weight Heparin Cotreatment, Alone and/or in Combination on Implantation and Clinical Pregnancy Rates in Repeated Implantation Failures in IVF Cycle.
Brief Title: Effects of Aspirin and Low Molecular Weight Heparin in IVF Outcome.
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Dr.Vandana Bansal (Other)
Responsible Party: Sponsor-Investigator, Dr.Vandana Bansal, Director & Consultant, Jeevan Jyoti Hospital
Organization: Jeevan Jyoti Hospital (Other)
Allocation: Randomized | Model: Factorial | Masking: Single | Purpose: Treatment
Other Study IDs: JJH2013
Record Dates: First submitted 2013-08-12; First posted 2013-08-16 (Estimated); Last update posted 2013-08-16 (Estimated); Status verified 2013-08

CONDITIONS: To Investigate the Effects of Low Dose Aspirin and Low Molecular Weight Heparin in IVF Out Come
Keywords: IVF failure, implantation rate, heparin & aspirin
MeSH Terms: interventions — Heparin, Low-Molecular-Weight; Aspirin; Heparin

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Low Molecular Weight Heparin (Active Comparator): Low molecular weight heparin, 2500 milli-International unit/day, subcutaneously
  Interventions: Drug: Low molecular weight heparin
- Low dose aspirin (Active Comparator): Low dose aspirin, 75mg/day, orally
  Interventions: Drug: Low dose aspirin
- Heparin & Aspirin (Active Comparator): Heparin (40 mg/day, subcutaneously) and aspirin (70 mg/day, orally)
  Interventions: Drug: Heparin & aspirin
- Sodium chloride (NaCl) (Placebo Comparator): Equivalent volume of NaCl 0.9%, subcutaneously
  Interventions: Other: NaCl

INTERVENTIONS:
Drug: Low molecular weight heparin — 2500 mIU/day, subcutaneously
  Other Names: LMWH
  Arms: Low Molecular Weight Heparin
Drug: Low dose aspirin — 75 mg/day, orally
  Other Names: Ecoaspirin
  Arms: Low dose aspirin
Drug: Heparin & aspirin — Aspirin (70 mg/day, orally) & heparin (40 mg/day, subcutaneously)
  Other Names: LMWH & Ecoaspirin
  Arms: Heparin & Aspirin
Other: NaCl — Equivalent volume of NaCl 0.9%, subcutaneously
  Arms: Sodium chloride (NaCl)

SUMMARY:
The purpose of the study is to determine whether low-dose aspirin and low molecular weight heparin improve the implantation and pregnancy rates in patients with repeated implantation failures in IVF cycle.

DETAILED DESCRIPTION:
The investigators hypothesize that cotreatment of low dose aspirin & low molecular weight heparin may improve implantation & clinical pregnancy rates.

ELIGIBILITY:
Inclusion Criteria:

* Aged between 19 to 35 years;
* Basal follicle-stimulating hormone (FSH) levels of ≤8 IU/l
* Body mass index (BMI) between 19 kg/m2 and 25 kg/m2
* Presence of both ovaries; ≥2 previous IVF failures
* Good quality embryos for transfer
* Endometrial thickness between 10 mm and 14 mm

Exclusion Criteria:

* Polycystic ovary syndrome
* Endometriosis

Ages: 19 Years to 35 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 400 (Estimated)
Dates: Start 2013-08; Primary Completion 2014-08 (Estimated); Study Completion 2014-12 (Estimated)

PRIMARY OUTCOMES:
Biological pregnancy test | 14 days

SECONDARY OUTCOMES:
Fetal heart/Gestational sac | 8 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Vandana Bansal, MS DGO PhD, Principal Investigator — Arpit Test Tube Baby Centre, Vandana Women's Hospital, Jeevan Jyoti Hospital & Research Centre
Locations (1):
- Arpit Test Tube Baby Centre, Jeevan Jyoti Hospital & Research Centre, Allahābād, Uttar Pradesh, India